CLINICAL TRIAL: NCT02278315
Title: Phase 1, Open-Label, Dose Escalation Study of I-131-CLR1404 in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Dose Escalation Study of I-131-CLR1404 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCL-14-002
Record Dates: First submitted 2014-10-22; First posted 2014-10-30 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Radiopharmaceutical; Therapy; Phase 1
MeSH Terms: conditions — Multiple Myeloma | interventions — CLR1404; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental): I-131-CLR1404 with or without concurrent dexamethasone
  Interventions: Drug: I-131-CLR1404; Drug: dexamethasone

INTERVENTIONS:
Drug: I-131-CLR1404 — Single IV dose of I-131-CLR1404, increased/decreased by cohort
  Other Names: 131I-CLR1404; 18-(p-[I-131]-iodophenyl)octadecyl phosphocholine; CLR 131
Drug: dexamethasone — 40 mg dexamethasone orally once weekly for up to 12 weeks
  Other Names: Decadron
Drug: I-131-CLR1404 — Multiple IV dose of I-131-CLR1404, increased/decreased by cohort
  Other Names: 131I-CLR1404; 18-(p-[I-131]-iodophenyl)octadecyl phosphocholine; CLR 131

SUMMARY:
The primary objective of the study is to determine the safety and tolerability of I-131-CLR1404 as a single or multiple dose, with and without concurrent weekly dexamethasone, in patients with relapsed or refractory multiple myeloma who have previously been treated with, or are intolerant of, an immunomodulator and a proteasome inhibitor.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is an incurable, monoclonal proliferation of plasma cells. Approximately 80,000 Americans are affected by MM with approximately 22,000 new cases diagnosed and 11,000 deaths each year. The introduction of newer therapies in the past twenty years, such as autologous stem cell transplantation and novel agents such as proteasome inhibitors and immune modulating drugs has improved outcomes, with current median overall survival estimates of 3-10 years depending on a number of patient-, disease- and treatment-related factors. However, despite these innovations, myeloma relapse is inevitable. Therefore, there is a clear need for improved therapies for MM and, in particular, for relapsed disease.

I-131-CLR1404 is a radioiodinated therapeutic that exploits the selective uptake and retention of phospholipid ethers (PLEs) by malignant cells. Cellectar Biosciences' novel cancer-targeted small-molecule compound (CLR1404) is radiolabeled with the isotope iodine-131 (I-131). Radioiodinated CLR1404 has been evaluated in over 60 xenograft and spontaneous (transgenic) tumor models. In all but two cases of hepatocellular carcinoma, CLR1404 demonstrated selective cancer cell uptake and retention. In various rodent tumor models, I-131-CLR1404 has also demonstrated tumor growth delay and prolongation of survival.

Based on the critical unmet medical need for effective agents with novel mechanisms of action in MM, the exquisite radiosensitivity of MM, and initial preclinical and clinical experience with radioiodinated CLR1404, Cellectar Biosciences has chosen to assess I-131-CLR1404 in a MM-specific phase 1 trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed multiple myeloma
* Prior treatment with or intolerance to proteasome inhibitor and immunomodulator
* Bone marrow biopsy within 28 days of study drug infusion demonstrating at least 5% plasma cell involvement
* Progressive disease defined by any of following:

  25% increase in serum M-protein from lowest response value during (or after) last therapy and/or absolute increase in serum M-protein of > or equal to 0.5 g/dL; 25% increase in urine M-protein from lowest response value during (or after) last therapy and/or absolute increase in urine M-protein of > or equal to 200 mg/24h; 25% increase in bone marrow plasma cell percentage from lowest response value during (or after) last therapy - absolute bone marrow plasma cell percentage must be > or equal to 10% unless prior complete response when absolute bone marrow plasma cell percentage must be > or equal to 5%; 25% increase in serum FLC level from the lowest response value during (or after) last therapy - the absolute increase must be > 10 mg/dL; new onset hypercalcemia > 11.5 mg/dL
* Measurable disease defined by any of following: Serum M-protein > 1 g/dL; Urine M-protein > 200 mg/24h; Serum free light chain (FLC) assay: involved FLC level > or equal to 10 mg/dL provided serum FLC ratio is abnormal; subjects who are non-secretors will be considered on a case-by-case basis
* Eastern Cooperative Oncology Group performance status of 0 to 2
* Life expectancy of at least 6 months
* Have initiative and means to be compliant with protocol and within geographical proximity to make required study visits as judged by Investigator
* Subject or legal representative has ability to read, understand and provide written informed consent for study related procedures
* Women of childbearing potential must have negative pregnancy test within 24 hours of enrollment
* Women of childbearing potential and men who are able to father a child, must agree to use an effective contraception method during study and for 12 months following study drug administration

Exclusion Criteria:

* Grade 2 or greater toxicities due to previous therapies, subject to laboratory abnormalities listed below. Stable, tolerable Grade 2 adverse events may be allowed at discretion of Investigator
* Prior external beam radiation therapy resulting in greater than 20% total bone marrow receiving greater than 20 Gy
* Prior radioisotope therapy
* Prior total body or hemi-body irradiation
* Extradural tumor in contact with the spinal cord or tumor located where swelling in response to therapy may impinge upon spinal cord
* Subject has any of following laboratory abnormalities: WBC < 3000/uL; ANC < 1500/uL; Hemoglobin < 8 g/dL; Estimated glomerular filtration rate < 30 mL/min/1.73 m2; ALT > 3 x ULN ; Bilirubin > 1.5 x ULN
* Platelet count < 100,000/uL without full-dose anticogulation therapy
* Platelet count < 150,000/uL with ongoing full-dose anticoagulation therapy
* Clinically significant bleeding event, as judged by investigator, within prior 6 months
* Chronic immunosuppressive therapy
* Anti-platelet therapy, except low-dose aspirin for cardioprotection
* PTT > 1.3 x ULN
* INR > 1.3
* Radiation therapy, chemotherapy, immunotherapy, investigational therapy or corticosteroid use within 2 weeks of or after eligibility-defining bone marrow biopsy. Bisphosphonates and denosumab are permitted if subject has been receiving for at least 90 days
* History of hypersensitivity to iodine
* Any other concomitant serious illness or organ system dysfunction in opinion of Investigator would either compromise subject safety or interfere with test drug safety evaluation
* Major surgery within 6 weeks of enrollment
* Known history of HIV, hepatitis C or hepatitis B infection
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLT) | up to 85 days
  DLT will be assessed by physical examination, vital signs, ECG, and laboratory values

SECONDARY OUTCOMES:
Identification of recommended phase 2 dose of I-131-CLR1404 with concurrent weekly dexamethasone | until non-tolerated dose is defined; dose escalation descision made upon review of data from a complete cohort (85 days after all subjects in cohort have received infusion)
  Largest administered dose with concurrent weekly dexamethasone with at most a 17% dose limiting toxicity rate
Identification of recommended phase 2 dose of I-131-CLR1404 without dexamethasone | until non-tolerated dose is defined; dose escalation descision made upon review of data from a complete cohort (85 days after all subjects in cohort have received infusion)
  Largest administered dose without dexamethasone with at most a 17% dose limiting toxicity rate
Identify the recommended dosing schedule of I-131-CLR1404, in relapsed or refractory MM | until non-tolerated dose is defined with both dosing regimens; dose escalation decision made upon review of data from a complete cohort (85 days after all subjects in cohort have received infusion)

OTHER OUTCOMES:
Determination of therapeutic activity of I-131-CLR1404 in relapsed or refractory multiple myeloma | through Day 85
  Response assessment per International Uniform Response Criteria for Multiple Myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Natalie S Callander, MD, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Mayo Clinic, Jacksonville, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Background] Weichert JP, Clark PA, Kandela IK, Vaccaro AM, Clarke W, Longino MA, Pinchuk AN, Farhoud M, Swanson KI, Floberg JM, Grudzinski J, Titz B, Traynor AM, Chen HE, Hall LT, Pazoles CJ, Pickhardt PJ, Kuo JS. Alkylphosphocholine analogs for broad-spectrum cancer imaging and therapy. Sci Transl Med. 2014 Jun 11;6(240):240ra75. doi: 10.1126/scitranslmed.3007646. PMID 24920661